CLINICAL TRIAL: NCT06198686
Title: An Evaluation of The Absolute Bioavailability of TH104
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tharimmune Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: TH104-105
Record Dates: First submitted 2023-12-27; First posted 2024-01-10 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Healthy
MeSH Terms: interventions — nalmefene

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental): A buccal formulation of Nalmefene 16 mg and a 1 mg intravenous dose of nalmefene injection, with a least 7 days washout period between dose
  Interventions: Drug: Nalmefene
- Sequence 2 (Experimental): A 1 mg intravenous dose of nalmefene injection, and a buccal formulation of Nalmefene 16 mg with a least 7 days washout period between dose
  Interventions: Drug: Nalmefene

INTERVENTIONS:
Drug: Nalmefene — Opioid antagonist

SUMMARY:
This is a single-dose, single-center, open-label, randomized, 2-way crossover study (2 treatments, 2 periods and 2 sequences) of a buccal formulation of Nalmefene 16 mg and a 1 mg intravenous dose of nalmefene injection, with a least 7 days washout period between doses.

ELIGIBILITY:
Inclusion Criteria:

1. Subject age between 18 to 55 years old.
2. Subject body weight ≤ 120 kg, with a BMI within of 18-30 kg/m2
3. Subject is able to complete the clinical study including the follow-up.
4. Subject is capable of providing written informed consent.

Exclusion Criteria:

1. Breastfeeding female.
2. Positive pregnancy test (female).
3. Systolic blood pressure outside 80-140 mm Hg or diastolic blood pressure outside 50-80 mm Hg.
4. Bradycardia defined as symptomatic heart rate < 60 bpm or asymptomatic heart rate < 55 bpm and tachycardia defined as resting heart rate > 100 bpm.
5. Clinically significant ECG abnormalities.
6. QTc > 450 ms for male and > 460 ms for female.
7. A history of allergies, or any significant adverse reactions, to any medications.
8. A history of seizures or convulsions.
9. Clinically significant medical, familial, or surgical history of eyes, ears, nose, throat, respiratory, cardiovascular, gastrointestinal, genitourinary, neurological, hematopoietic, lymphatic, endocrine, metabolic, dermatological, musculoskeletal, psychological and/or other major disease or malignancy.
10. Family history of sudden cardiac death.
11. Clinically significant physical examination finding.
12. Clinically significant laboratory abnormalities.
13. Hemoglobin < 12.0 g/dL for male and < 11.0 g/dL for female at screening.
14. Creatinine clearance <90 mL/m2/min
15. Total bilirubin , ALT/AST greater than upper limit of normal, or CPK > 2 x upper limit of normal.
16. Hepatitis B, Hepatitis C or HIV positive.
17. Positive test for drugs of abuse.
18. Smoke more than 10 sticks of cigarettes a day, vape more than 20 mg of liquid nicotine a day, or equivalent.
19. A history of drug or substance abuse, including alcohol (≥ 7 units per week) within 6 months before dosing (1 unit of alcohol equals approximately ½ pint [240 mL] of beer, 1 glass [125 mL] of wine, or 1 shot [25 mL] of spirit).
20. Have taken any medications (including herbal remedies) within 7 days before dosing, with the exception of birth control medications and other medications deemed acceptable by the Investigator.
21. Use of any opioid antagonist (e.g., naloxone, naltrexone, nalmefene) in the past.
22. Clinically significant illness or injury or hospitalization for any reason within 28 days before dosing.
23. Participation in other clinical study involving a marketed or investigational drug within 28 days or 10 half-lives of the drug before dosing, whichever is longer.
24. Donation of > 500 mL of plasma within 14 days before dosing; or donation or loss of whole blood (excluding the amount of blood collected during screening) before dosing as follows:

    * 50-300 mL within 28 days,
    * 301-500 mL within 42 days, or
    * 500 mL within 84 days.
25. Any other medical condition or reason that, in the opinion of the Investigator or Research Physician, makes the subject unsuitable to participate in the clinical study.
26. Female of childbearing potential having unprotected sexual intercourse with any non-sterile male partner within 14 days before dosing and until 60 days after receiving the last dose; acceptable methods of contraception include:

    * double barrier (1 by each partner), and at least 1 of these barriers (condom, cervical cap, diaphragm or sponge) must contain spermicide,
    * hormonal (oral, injectable, transdermal, intravaginal or implantable),
    * intrauterine contraceptive system,
    * surgical (vasectomy or tubal ligation), or
    * sexual abstinence.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-01-26 (Actual); Primary Completion 2024-02-11 (Actual); Study Completion 2024-11-06 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration Versus Time Curve (AUC) of Nalmefene | 4 days
  Determine the absolute bioavailability of a buccal dose of TH104

SECONDARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events | 4 days
  To compare the tolerability of TH104 films with intravenous nalmefene

CONTACTS AND LOCATIONS:
Locations (1):
- Novum Pharmaceutical Research Services, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No